CLINICAL TRIAL: NCT05962879
Title: Development of a Transdiagnostic Intervention for Adolescents at Risk for Serious Mental Illness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Nicole DeTore, PhD, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023P000985; K23MH131793 (NIH)
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Anxiety Disorders; Psychotic Disorders; Depressive Disorder; Psychosocial Functioning
MeSH Terms: conditions — Anxiety Disorders; Psychotic Disorders; Depressive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resilience Training for Teens (Experimental): A brief 6-session group-based behavioral intervention for teens at risk of a mental illness.
  Interventions: Behavioral: Resilience Training for Teens
- Waitlist (No Intervention): A one year waitlist period where participants will not participate in Resilience Training for Teens. Following that one year waitlist period, they can participate in Resilience Training for Teens.

INTERVENTIONS:
Behavioral: Resilience Training for Teens — A brief 6-session group-based behavioral intervention for high school aged teenagers at risk of a mental illness.
  Arms: Resilience Training for Teens

SUMMARY:
This research study aims to develop a brief group-based treatment called Resilience Training for Teens, then to test how well it protects high school students with mild symptoms of depression, anxiety, or having unusual feelings from developing mental illnesses.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in 9th through 12th grade and between the ages of 14 and 19
* Endorsed at least one psychotic experience
* Provided contact information
* Have a parent or legal guardian who is able and willing to provide written informed consent (if under the age of 18)
* Have a parent or legal guardian who is able and willing to participate in a parent session
* Competent and willing to provide written informed assent (if under the age of 18) or consent (if age 18 or older)
* Able to communicate in English

Exclusion Criteria:

* Currently prescribed psychotropic medication (not including medications for attention deficit/hyperactivity disorder), regardless of adherence
* Currently obtaining psychotherapeutic intervention

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Structured Interview of Psychosis-risk Syndromes (SIPS) | 1 year
  Subclinical psychotic symptoms that represent a risk of transdiagnostic mental illnesses. This semi-structured interview rates psychotic experiences, general symptoms, and functioning. The SIPS interview assesses positive, negative, disorganized, and general symptoms. The range of the Scale of Psychosis-risk Symptoms (SOPS) is 0-6, with a higher score representing more severe symptoms.

SECONDARY OUTCOMES:
Child Behavior Checklist (CBCL) | 1 year
  Mental health symptoms in the teen rated by both the teen and the parent/guardian consisting of 113 items. The CBCL rates multiple domains across functioning and psychiatric diagnoses. It is scored on a 3-point Likert scale, with higher scores representing more severe symptoms.
Global Functioning Social and Role Scales | 1 year
  Social and school/work functioning captured on this scale rated on a 10 point likert scale assessing functional and social functioning separately. Higher ratings represent richer functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided